CLINICAL TRIAL: NCT05361655
Title: Real-World Treatment Effectiveness of Palbociclib in Combination With an Aromatase Inhibitor as 1st Line Therapy in Metastatic Breast Cancer
Brief Title: Real-World Effectiveness of Palbociclib in Combination With an Aromatase Inhibitor
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481151
Record Dates: First submitted 2022-04-21; First posted 2022-05-05 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Breast Cancer
Keywords: cyclin-dependent kinase 4/6i (CDK4/6i)
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Palbociclib + an aromatase inhibitor: Adult metastatic breast cancer patients who initiated Palbociclib + an aromatase inhibitor as first line therapy between Feb 3, 2015 to March 31, 2020 in the Flatiron Health Analytic Database.
  Interventions: Drug: Palbociclib + an aromatase inhibitor
- Aromatase inhibitor: Adult metastatic breast cancer patients who initiated an aromatase inhibitor as first line therapy between Feb 3, 2015 to March 31, 2020 in the Flatiron Health Analytic Database.
  Interventions: Drug: Aromatase inhibitor

INTERVENTIONS:
Drug: Palbociclib + an aromatase inhibitor — Palbociclib + an aromatase inhibitor therapy
  Groups: Palbociclib + an aromatase inhibitor
Drug: Aromatase inhibitor — Aromatase inhibitor therapy
  Groups: Aromatase inhibitor

SUMMARY:
A retrospective study of de-identified (to preserve patient privacy) patient information from the Flatiron Health Analytic Database to compare effectiveness (i.e., overall survival) of first line palbociclib + aromatase inhibitor (AI) versus AI alone treatment in postmenopausal women or men with hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-) metastatic breast cancer (MBC) in the United States clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HR+/HER2- status after MBC diagnosis.
* Received palbociclib + AI or AI as first-line therapy

Exclusion Criteria:

* Evidence of prior treatment with other CDK4/6I, AI, tamoxifen, raloxifene, toremifene, or Fulvestrant for MBC
* First structured activity greater than 90 days after MBC diagnostic date
* Treatment with a CDK4/6 inhibitor as part of a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+/HER2- MBC adult patients treated with Palbociclib + AI or AI alone between February2015 and September, 2020
Sampling Method: Non-Probability Sample
Enrollment: 2888 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- 10017, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Layman RM, Liu X, Li B, McRoy L, Brufsky A. Real-world palbociclib dose modifications and clinical outcomes in patients with HR+/HER2- metastatic breast cancer: A Flatiron Health database analysis. Breast. 2025 Jun;81:104448. doi: 10.1016/j.breast.2025.104448. Epub 2025 Mar 17. PMID 40138984
- [Derived] Brufsky A, Liu X, Li B, McRoy L, Chen C, Makari D, Layman RM, Rugo HS. Palbociclib plus aromatase inhibitors in patients with metastatic breast cancer and cardiovascular diseases: real-world effectiveness. Oncologist. 2024 Dec 6;29(12):1032-1043. doi: 10.1093/oncolo/oyae273. PMID 39418346
- [Derived] Rugo HS, Liu X, Li B, McRoy L, Chen C, Layman RM, Tomlin-Harris T, Brufsky A. Prolonging the lives of African-Americans with metastatic breast cancer by adding palbociclib to an aromatase inhibitor in routine clinical practice: a plain language summary of a real-world database study. Future Oncol. 2024;20(19):1299-1307. doi: 10.2217/fon-2023-1079. Epub 2024 Mar 22. PMID 38517416
- [Derived] Rugo HS, Liu X, Li B, McRoy L, Chen C, Layman RM, Brufsky A. Real-World Effectiveness of Palbociclib Plus Aromatase Inhibitors in African American Patients With Metastatic Breast Cancer. Oncologist. 2023 Oct 3;28(10):866-874. doi: 10.1093/oncolo/oyad209. PMID 37487056
- [Derived] Rugo HS, Brufsky A, Liu X, Li B, McRoy L, Chen C, Layman RM, Cristofanilli M, Torres MA, Curigliano G, Finn RS, DeMichele A. Prolonging the life of people with metastatic breast cancer in routine clinical practice by adding palbociclib to an aromatase inhibitor from a real-world database analysis: a plain language summary. Future Oncol. 2023 Mar;19(7):489-498. doi: 10.2217/fon-2022-1192. Epub 2023 Mar 9. PMID 36892508
- [Derived] Rugo HS, Brufsky A, Liu X, Li B, McRoy L, Chen C, Layman RM, Cristofanilli M, Torres MA, Curigliano G, Finn RS, DeMichele A. Real-world study of overall survival with palbociclib plus aromatase inhibitor in HR+/HER2- metastatic breast cancer. NPJ Breast Cancer. 2022 Oct 11;8(1):114. doi: 10.1038/s41523-022-00479-x. PMID 36220852
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women or men with human epidermal growth factor receptor positive(HR+)/human epidermal growth factor receptor 2 negative(HER2-)metastatic breast cancer(MBC)who initiated first line treatment with palbociclib + aromatase inhibitor(AI)or AI alone from February 2015 through March 2020 and were registered in the Flatiron Health Analytic Database were included in the study. Participants were followed until death or study end (date of data cutoff, 30-Sep-2020), whichever occurred first.
Pre-assignment Details: All participants who were eligible for the retrospective database analysis were included for the study (i.e., 2888).
Groups:
- Palbociclib + Aromatase Inhibitor: Participants with HR+/HER2- MBC who initiated first line treatment with palbociclib + aromatase inhibitor between 03 Feb 2015 to 31 Mar 2020 were included and observed.
- Aromatase Inhibitor: Participants with HR+/HER2- MBC who initiated first line treatment with aromatase inhibitor alone between 03 Feb 2015 to March 2020 were included and observed.
Period: Overall Study
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Started | 1324 | 1564
Completed | 1324 | 1564
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population comprised of all eligible participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor | Total
Number analyzed (Participants) | 1324 | 1564 | 2888
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 516 | 416 | 932
  >=65 years | 808 | 1148 | 1956
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1314 | 1545 | 2859
  Male | 10 | 19 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 900 | 1059 | 1959
  Black | 107 | 136 | 243
  Unknown | 317 | 369 | 686

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Postmenopausal Female or Male Participants With Metastatic Breast Cancer
Description: OS was defined as the time from the index date (start of palbociclib + AI or AI alone) to death. Participants who did not die, were censored at the end of study date (30-Sep-2020). Kaplan-Meier method adjusted by stabilized inverse probability of treatment weighting (sIPTW) was used.
Time Frame: From index date to death due to any cause or censoring date of 30-Sep-2020 (approximately up to 68 months)
Population: FAS population comprised of all eligible participants enrolled in the study. Analysis was performed using sIPTW method to balance participant characteristics among reporting groups. sIPTW method created balanced virtual groups and hence overall number of participants analyzed was different from numbers in participant flow (not balanced).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1572 | 1137
Months | 49.1 [45.2 to 57.7] | 43.2 [37.6 to 48.0]
Statistical Analysis 1: Comparison: Palbociclib + Aromatase Inhibitor vs Aromatase Inhibitor; Test type: Other; p < 0.0001, Cox proportional hazard model; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.65 to 0.87]

2. Secondary Outcome: Real-World Progression Free Survival (rwPFS) in Postmenopausal Female or in Male Participants With Metastatic Breast Cancer
Description: Real-world PFS was defined as the number of months from start of palbociclib + AI or AI alone to death from any cause or disease progression (based on clinical assessment or by radiographic scan/tissue biopsy), whichever occurred first. Disease progression was defined as at least a 20 percentage (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that was the smallest on study). Participants who did not die and did not have disease progression were censored at the date of initiation of next line of therapy for participants with 2 or more lines of therapy or at the date of their last visit during the study period (February 2015-September 2020) for participants with only 1 line of therapy. Kaplan-Meier method adjusted by stabilized IPTW was used.
Time Frame: From index date until disease progression or death due to any cause or censoring date (approximately up to 68 months)
Population: FAS population comprised of all eligible participants enrolled in the study. Analysis was performed using sIPTW method to balance participant characteristics among reporting groups. sIPTW method created balanced virtual groups and hence overall number of participants analyzed was different from numbers in participant flow(not balanced).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1572 | 1137
Months | 19.3 [17.5 to 20.7] | 13.9 [12.5 to 15.2]
Statistical Analysis 1: Comparison: Palbociclib + Aromatase Inhibitor vs Aromatase Inhibitor; Test type: Other; p < 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.62 to 0.76]

3. Secondary Outcome: Number of Participants According to Real-World Tumor Responses (rwTR): Postmenopausal Female or in Male Participants With Metastatic Breast Cancer
Description: Real-world best responses were assessed based on treating clinician's assessment of radiological evidence for change in burden of disease over course of treatment after 1 month of index treatment initiation. Responses were classified as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), indeterminate response (IR). CR=Complete resolution of all visible disease. PR=partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. SD=no change in overall size of visible disease. PD: an increase in visible disease; also included cases where some lesions increased in size and some lesions decreased in size; included cases where clinician indicated progressive disease; IR=study data not available for evaluation of efficacy for any reason, including participants lost to follow-up or assessment not undertaken or death. Analysis was performed using sIPTW method to balance participant characteristics.
Time Frame: From 30 days after index treatment initiation until CR, PR, SD or PD (approximately 67 months)
Population: FAS population comprised of all eligible participants enrolled in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1263 | 988
Participants
  Complete response | 163 | 86
  Partial response | 569 | 300
  Stable disease | 350 | 273
  Progressive disease | 155 | 260
  Indeterminate response | 26 | 69

4. Secondary Outcome: Real-World Response Rate (rwTR) in Postmenopausal Female or in Male Participants With Metastatic Breast Cancer
Description: Real-world tumor response rate (rwTR) was defined as the percentage of participants with a real world complete response (rwCR) or real-world partial response (rwPR). CR: complete resolution of all visible disease. PR: partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. Analysis was performed using sIPTW method to balance participant characteristics.
Time Frame: From 30 days after index treatment initiation until disease progression or death due to any cause or censoring date (approximately up to 67 months)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1263 | 988
Percentage of participants | 57.98 | 39.04
Statistical Analysis 1: Comparison: Palbociclib + Aromatase Inhibitor vs Aromatase Inhibitor; Test type: Other; p < 0.0001, score test

5. Secondary Outcome: Number of Participants According to Initial Dose of Palbociclib: Palbociclib + Aromatase Inhibitor Arm Only
Description: Number of participants according to the initial dose of palbociclib (75 milligrams [mg]/day, 100mg/day, 125 mg/day or missing dose) are reported in this outcome measure.
Time Frame: At index (anytime between 03-Feb-2015 to 31-Mar-2020, approximately up to 62 months)
Population: FAS population comprised of all eligible participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Aromatase Inhibitor
Number analyzed (Participants) | 1324
Participants
  Palbociclib 75 mg/day | 48
  Palbociclib 125 mg/day | 1110
  Palbociclib 100 mg/day | 144
  Missing | 22

6. Secondary Outcome: Time to Dose Adjustment for Palbociclib- Palbociclib + Aromatase Inhibitor Arm Only
Description: Time to dose adjustment for participants who received palbociclib 125 mg/day, 100 mg/day, or 75 mg/day as initial dose was presented in this outcome measure.
Time Frame: At index (anytime between 03-Feb-2015 to 30-Sep-2020, approximately up to 68 months)
Population: FAS population comprised of all eligible participants enrolled in the study. Here 'Overall Number of Participants Analyzed' signifies the total number of participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Palbociclib + Aromatase Inhibitor
Number analyzed (Participants) | 1302
Days
  Initial dose of 125mg/day: number analyzed (Participants) | 1110
  Initial dose of 125mg/day | 85 [52 to 195]
  Initial dose of 100mg/day: number analyzed (Participants) | 144
  Initial dose of 100mg/day | 95 [39 to 236]
  Initial dose of 75mg/day: number analyzed (Participants) | 48
  Initial dose of 75mg/day | 112 [39 to 171]

7. Secondary Outcome: Duration of Treatment
Description: Duration of treatment was defined as days from index prescription order date to end of treatment, start of subsequent line of therapy, or death from any cause, whichever occurred first. Kaplan-Meier method adjusted by stabilized IPTW was used.
Time Frame: From start of study treatment to end of treatment, start of subsequent line of therapy, or death from any cause, whichever occurred first (up to 68 months)
Population: FAS population comprised of all eligible participants enrolled in the study. sIPTW method created balanced virtual groups and hence overall number of participants analyzed was different from numbers in participant flow (not balanced).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1572 | 1137
Months | 12.3 [10.5 to 14.1] | 5.5 [4.7 to 6.7]
Statistical Analysis 1: Comparison: Palbociclib + Aromatase Inhibitor vs Aromatase Inhibitor; Test type: Other; p < 0.0001, Cox proportional hazard model; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.60 to 0.72]

8. Secondary Outcome: Time to Next Line of Treatment
Description: Time to next line of treatment represents the interval from commencement of one treatment to initiation of the next line of therapy. Analysis was performed using sIPTW method to balance participant characteristics among reporting groups.
Time Frame: From start of study treatment to start of next line of therapy (up to 68 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1572 | 1137
Months | 18.4 [16.3 to 20.3] | 8.3 [7.2 to 10.2]
Statistical Analysis 1: Comparison: Palbociclib + Aromatase Inhibitor vs Aromatase Inhibitor; Test type: Other; p < 0.0001, Cox proportional hazard model; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.51 to 0.62]

9. Secondary Outcome: Time to Subsequent Chemotherapy
Description: Time to subsequent chemotherapy represents the time interval to administration of a different chemotherapeutic agent after the first course of therapy was administered. Analysis was performed using sIPTW method to balance participant characteristics among reporting groups.
Time Frame: From start of study treatment to administration of different chemotherapeutic agent (up to 68 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1572 | 1137
Months | 37.4 [33.7 to 40.7] | 29.2 [26.8 to 33.5]
Statistical Analysis 1: Comparison: Palbociclib + Aromatase Inhibitor vs Aromatase Inhibitor; Test type: Other; p < 0.0001, Cox proportional hazard model; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.69 to 0.86]

10. Secondary Outcome: Real-World Progression Free Survival 2 (rwPFS2) in Postmenopausal Female or in Male Participants With Metastatic Breast Cancer
Description: rwPFS2 was defined as the time from the index date to the date of the first documentation of a rwPD or death due to any cause after starting second line of therapy, whichever occurs first. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Analysis was performed using sIPTW method to balance participant characteristics among reporting groups.
Time Frame: From start of study treatment until disease progression, or death from any cause following second line of therapy, whichever occurred first (approximately up to 68 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
Number analyzed (Participants) | 1572 | 1137
Months | 32.6 [29.4 to 35.2] | 20.7 [18.9 to 22.6]
Statistical Analysis 1: Comparison: Palbociclib + Aromatase Inhibitor vs Aromatase Inhibitor; Test type: Other; p < 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.54 to 0.70]

ADVERSE EVENTS:
Time Frame: Overall survival: An outcome measures in the study, estimated from index date to death due to any cause or end of study (up to 68 months). However, in the retrospective deidentified database analysis, individual identifying information, cause of death, and data for non-serious adverse events and serious adverse events (SAEs) were not available and hence were not evaluated during the study.
Description: In this observational retrospective study of deidentified database individual identifying information was not available. Minimum criteria for reporting an adverse event could not be met, hence SAEs and other AEs were not planned to be collected and reported.
Arm/Group | Palbociclib + Aromatase Inhibitor | Aromatase Inhibitor
All-Cause Mortality (participants affected / at risk) | 420/1324 | 736/1564
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT05361655/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT05361655/SAP_001.pdf